CLINICAL TRIAL: NCT04497766
Title: Comparasion of Efficacy of Nebulized Magnesium Sulphate With Intravenous Magnesium Sulphate in Children With Acute Asthma
Brief Title: Comparasion of Efficacy of Nebulized With Intravenous Magnesium Sulphate in Children With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saima Khatoon (Other)
Collaborators: King Edward Medical University (Other)
Responsible Party: Sponsor-Investigator, Saima Khatoon, Post Graduate Resident in Pediatrics (MD Paeds), King Edward Medical University
Organization: King Edward Medical University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 137/RC/KEMU
Record Dates: First submitted 2020-07-16; First posted 2020-08-04 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Asthma in Children
Keywords: asthma in children; intravenous magnesium sulphate; nebulized magnesium sulphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebulized magnesium sulphate (Experimental): 100mg of mgso4 in 20ml of normal saline via ultrasonic nebulizer
  Interventions: Drug: Nebulized Magnesium sulfate
- Intravenous magnesium sulphate (Experimental): Magnesium sulphate according to weight will be given intravenously.
  Interventions: Drug: Intravenous magnesium sulphate

INTERVENTIONS:
Drug: Nebulized Magnesium sulfate — MgSO4 100mg in 20 ml normal saline will be given via ultrasonic nebulizer over 10 minutes,and PAS score will be assessed at 30,60,120,240,360 minutes
  Other Names: Nebulized MgSO4
  Arms: Nebulized magnesium sulphate
Drug: Intravenous magnesium sulphate — pts age 2 to 12 years will receive intravenous magnesium sulphate 50 mg/kg over half hour
  Other Names: IV MgSO4
  Arms: Intravenous magnesium sulphate

SUMMARY:
The purpose of study is to assess the effectiveness of nebulized magnesium sulphate in children presenting with acute asthma.Study perfoma consists of demographic variables,exclusion criteria and pediatric asthma score that includes respiratory rate,SPO2 at room air(requirement of oxygen),auscultatory findings in chest,dysnea and retractions.

DETAILED DESCRIPTION:
After getting informed consent from guardian,148 patients of acute moderate ro severe asthma with pediatric asthma score 8-15 will be randomly classified into 2 groups and one group will receive nebulization with magnesium sulphate and other will receive intravenous magnesium sulphate and effectiveness will be compared by 4 point reduction in PAS from baseline in either groups after 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* patients with age 2 to 12 years with acute moderate to severe exacerbation of asthma as per operational definition children who are unrespoinsive to standard treatment of asthma at 60 minutes

Exclusion Criteria:

* those with history of chronic lung disease and abnormal renal function contraindication for MgSO4 due to hepatic or renal disease allergy to MgSo4 children who has other comorbid illness

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of nebulized magnesium sulphate with intravenous magnesium sulphate in children with acute asthma will be assessed by a drop in PAS score, as assessed at 6 hours of intervention. | 6 hours
  The intervention will be considered effective if there is a drop of at least 4 points in PAS score at hour-6 of intervention.

SECONDARY OUTCOMES:
duration of ICU stay | 72 hours/3 days
  this will be measured in hours
duration of hospital stay | 120 hours/5 days
  this will be measured in hours

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad-Haroon Hamid, MBBS,FCPS,FRCP, Principal Investigator — chairman /Head of department of pediatrics unit1 K.E medical university/mayo hospital l
Locations (1):
- King edward medical university/mayo hospital lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data will be shared after publication on a reasonable request.

REFERENCES:
- [Background] Powell C, Kolamunnage-Dona R, Lowe J, Boland A, Petrou S, Doull I, Hood K, Williamson P; MAGNETIC study group. Magnesium sulphate in acute severe asthma in children (MAGNETIC): a randomised, placebo-controlled trial. Lancet Respir Med. 2013 Jun;1(4):301-8. doi: 10.1016/S2213-2600(13)70037-7. Epub 2013 Apr 22. PMID 24429155
- [Background] Kokotajlo S, Degnan L, Meyers R, Siu A, Robinson C. Use of intravenous magnesium sulfate for the treatment of an acute asthma exacerbation in pediatric patients. J Pediatr Pharmacol Ther. 2014 Apr;19(2):91-7. doi: 10.5863/1551-6776-19.2.91. PMID 25024668
- [Background] Goodacre S, Cohen J, Bradburn M, Gray A, Benger J, Coats T; 3Mg Research Team. Intravenous or nebulised magnesium sulphate versus standard therapy for severe acute asthma (3Mg trial): a double-blind, randomised controlled trial. Lancet Respir Med. 2013 Jun;1(4):293-300. doi: 10.1016/S2213-2600(13)70070-5. Epub 2013 May 17. PMID 24429154
- [Background] Singhi S, Grover S, Bansal A, Chopra K. Randomised comparison of intravenous magnesium sulphate, terbutaline and aminophylline for children with acute severe asthma. Acta Paediatr. 2014 Dec;103(12):1301-6. doi: 10.1111/apa.12780. Epub 2014 Oct 2. PMID 25164315
- [Background] Shan Z, Rong Y, Yang W, Wang D, Yao P, Xie J, Liu L. Intravenous and nebulized magnesium sulfate for treating acute asthma in adults and children: a systematic review and meta-analysis. Respir Med. 2013 Mar;107(3):321-30. doi: 10.1016/j.rmed.2012.12.001. Epub 2013 Jan 3. PMID 23290189
- [Background] Alansari K, Ahmed W, Davidson BL, Alamri M, Zakaria I, Alrifaai M. Nebulized magnesium for moderate and severe pediatric asthma: A randomized trial. Pediatr Pulmonol. 2015 Dec;50(12):1191-9. doi: 10.1002/ppul.23158. Epub 2015 Feb 4. PMID 25652104
- [Background] Albuali WH. The use of intravenous and inhaled magnesium sulphate in management of children with bronchial asthma. J Matern Fetal Neonatal Med. 2014 Nov;27(17):1809-15. doi: 10.3109/14767058.2013.876620. Epub 2014 Jan 30. PMID 24345031
- [Background] Daengsuwan T, Watanatham S. A comparative pilot study of the efficacy and safety of nebulized magnesium sulfate and intravenous magnesium sulfate in children with severe acute asthma. Asian Pac J Allergy Immunol. 2017 Jun;35(2):108-112. doi: 10.12932/AP0780. PMID 27996280
- See also: Powell C, Dona RK, Lowe, J, Boland A, Petrou S, Doull I, et al. Magnesium sulphate in acute sever asthma in children (MAGNETIC): a randomized, placebo-controlled trial. The Lancet Respiratory Medicine. 2013;1(4):301-8. — http://pubmed.ncbi.nlm.nih.gov/24429155/
- See also: Kokotajlo S, Degnan L, Meyers R, Siu A, Robinson C. Use of intravenous magnesium sulfate for the treatment of an acute asthma exacerbation in pediatric patients.J Pediatr Pharmacol Ther. 2014;19(2) :91-7. — https://pubmed.ncbi.nlm.nih.gov/25024668
- See also: Goodacre S, Cohen J, Research Team. Intravenous or nebulised magnesium sulphate versus standard therapy for severe acute asthma (3Mg trial): a double-blind, randomised controlled trial.Lancet Respir Med. 2013;1(4 — http://pubmed.ncbi.nlm.nih.gov/24429154/
- See also: Singhi S, Grover S, Bansal A, Chopra K. Randomised comparison of intravenous magnesium sulphate, terbutaline and aminophylline for children with acute severe asthma. Acta Peadiatrica. 2014;103(12):1301-6 — http://pubmed.ncbi.nlm.nih.gov/25164315/
- See also: Shan Z, Rong Y, Yang W, Wang D, Yao P, Xie J,et al. Intravenous and nebulized magnesium sulfate for treating acute asthma in adults and children: a systematic review and meta-analysis. Respiratory medicine. 2013;107(3):321-30. — http://pubmed.ncbi.nlm.nih.gov/23290189/
- See also: Alansari K, Ahmed W, Davidson B, Alamri M, Zakaria I, Alrifaari M. Nebulized magnesium for moderate and severe pediatric asthma: A randomized tria.Pediatr Pumonol 2015;50(12):1191-9. — http://pubmed.ncbi.nlm.nih.gov/25652104/
- See also: Albuali WH. The Use of Intravenous and inhaled magnesium sulphate in management of children with bronchial asthma. J Matern Fetal Neonatal.2014;27(17):1809-15. — http://pubmed.ncbi.nlm.nih.gov/24345031/
- See also: aengsuwan T, Watanatham S. A comparative pilot study of the efficacy and safety of nebulized magnesium sulfate and intravenous magnesium sulfate in children with severe acute asthma. Asian Pac/allergy immunol. 2016; 35(2):108- — http://pubmed.ncbi.nlm.nih.gov/27996280/